CLINICAL TRIAL: NCT00449111
Title: An Open Label Study to Assess the Efficacy, Safety and Tolerability of COZAAR Plus (Losartan Potassium 50mg/Hydrochlorothiazide 12.5mg) Possibly Titrated up to COZAAR Plus-F (Losartan Potassium 100mg/Hydrochlorothiazide 25mg) in Patients With Essential Hypertension
Brief Title: An Open Label Study to Assess the Efficacy, Safety and Tolerability of COZAAR Plus (Losartan Potassium 50mg/Hydrochlorothiazide 12.5mg) Possibly Titrated up to COZAAR Plus-F (Losartan Potassium 100mg/Hydrochlorothiazide 25mg) in Patients With Essential Hypertension (0954A-325)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0954A-325; 2007_005
Record Dates: First submitted 2007-03-16; First posted 2007-03-19 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Losartan; Duration of Therapy

INTERVENTIONS:
Drug: MK0954, losartan potassium / Duration of Treatment - 12 weeks

SUMMARY:
Evaluate blood pressure after 6 weeks of treatment with COZAAR plus.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated with valsartan 80mg or irbesartan 150mg or vandesartan 8mg for at least 4 weeks prior to visit 1
* Patient with systolic blood pressure between 140 to 159 mmhg and diastolic pressure between 90 to 99mmhg taken at visit 1

Exclusion Criteria:

* History of angina pectoris that has not been stabilized in the past 6 weeks
* History of clinically significant abnormal lab results or diseases
* Myocardial infarction within the past 6 months
* Stroke in the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-03-13 (Actual); Primary Completion 2006-09-30 (Actual); Study Completion 2006-09-30 (Actual)

PRIMARY OUTCOMES:
Change of diastolic blood pressure after 6 weeks of treatment with cozaar plus

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC